CLINICAL TRIAL: NCT07103668
Title: An Open-label, Randomized, Comparative Phase III Study Including Patients With CLDN18.2-positive Unresectable Locally Advanced Gastric Cancer.
Brief Title: A Phase III Randomized Study in CLDN18.2-positive Unresectable Locally Advanced Gastric Cancer Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Immunofoco Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMC002-RT02-RCT
Record Dates: First submitted 2025-07-17; First posted 2025-08-05 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-08

CONDITIONS: Gastric Adenocarcinoma
MeSH Terms: interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IMC 002 CAR-T Cell Group (Experimental)
  Interventions: Drug: CAR T cells
- The anti-tumor drug selected by investigator (Active Comparator)
  Interventions: Drug: Control

INTERVENTIONS:
Drug: CAR T cells — better PFS/OS data comparing to the other studies.
  Arms: IMC 002 CAR-T Cell Group
Drug: Control — Chemo therapy by PI options.
  Arms: The anti-tumor drug selected by investigator

SUMMARY:
An open-label, randomized, comparative phase II study including patients with CLDN18.2-positive unresectable locally advanced gastric cancer. To evaluate the objective response rate (ORR) and progression-free survival (PFS) of IMC002 compared with investigator's choice of treatment (ICT) as third-line or later therapy in patients with unresectable locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma with positive CLDN18.2 expression.

ELIGIBILITY:
Inclusion Criteria:

1. The age at randomization was at least 18 years old , and both men and women were eligible.
2. histologically or cytologically confirmed inoperable locally advanced or metastatic gastric/esophagogastric junction adenocarcinoma who have failed at least two prior lines of therapy :

   1. Radiographic progression or clinical worsening of symptoms during second-line treatment (if first-line treatment includes three drugs including taxanes (or anthracyclines), platinums, and fluorouracils, and the disease progression is assessed by the investigator, the patient may also be enrolled as an eligible subject; disease progression within 6 months after the end of neoadjuvant/adjuvant treatment is also considered a first-line treatment failure);
   2. Patients with intolerance to second-line treatment may also be enrolled in the study after full evaluation by the investigator. The definition of intolerance to previous treatment is as follows:

   any Grade ≥ 3 (according to NCI CTCAE v5.0 criteria) hematologic toxicity that has not recovered to Grade 1 or pre-treatment levels after 14 days of best supportive care; any Grade ≥ 3 (according to NCI CTCAE v5.0 criteria) non-hematologic toxicity (excluding alopecia and asymptomatic laboratory abnormalities) that has not resolved after 14 days of best supportive care.
3. Tumor tissue specimens (primary or metastatic, archived or newly collected) from subjects are expected to be available and tested by a central laboratory, indicating positive histological staining for CLDN18.2 (defined as a positive tumor cell rate ≥40% and a staining intensity ≥2+) . If the subject has previously received other CLDN18.2-targeted therapies, tumor tissue specimens collected after that treatment are required to retest and evaluate CLDN18.2 expression levels .
4. The subject's expected survival period is ≥12 weeks.
5. According to RECIST 1.1, there should be at least one stably measurable target lesion or evaluable lesion, and the longest diameter of the largest lesion (or the shortest diameter if it is a lymph node lesion) should be ≤5 cm .
6. ECOG performance status score is 0-1.
7. The subject must have adequate organ and bone marrow function. Laboratory screening must meet the following criteria. All laboratory test results should be within the stable ranges described below, and there should be no ongoing supportive treatment. If any laboratory test result is abnormal based on the following criteria , the test can be repeated within 1 week. If the test results still do not meet the following criteria , the patient has failed the screening.

   1. Blood tests [no enhanced blood transfusion ( ≥ 2 times within 1 week), platelet transfusion, or cell growth factor (except recombinant erythropoietin) within 7 days before the examination]: neutrophil count ≥ 1.5×10 9 /L; platelet count (PLT) ≥ 75×10 9 /L; hemoglobin content (Hb) ≥ 8.0 g/dL; lymphocyte (LYM) ≥ 0.5×10 9 /L;
   2. Liver function: alanine aminotransferase (ALT) ≤ 2.5×ULN, aspartate aminotransferase (AST) ≤ 2.5×ULN, serum total bilirubin (TB) ≤ 2×ULN; for patients with liver metastasis, AST and ALT < 5×ULN;
   3. Renal function: Serum creatinine ≤ 1.5 × ULN. If serum creatinine is > 1.5 × ULN, creatinine clearance > 50 mL/min (based on the Cockcroft-Gault formula); qualitative urine protein ≤ 1+; if qualitative urine protein is ≥ 2+, a 24-hour urine protein quantitative test is required (a 24-hour urine protein quantitative test < 1 g is acceptable);
   4. Amylase and lipase ≤ 1.5 × ULN; alkaline phosphatase (ALP) ≤ 2.5 × ULN. For patients with bone metastases, ALP < 5 × ULN.
8. All toxic reactions caused by previous anti-tumor therapy have been alleviated to Grade 0-1 (according to NCI CTCAE Version 5.0) or to a level acceptable to the inclusion/exclusion criteria. This excludes other toxicities such as alopecia and vitiligo that the investigator believes do not pose a safety risk to the subjects.
9. Reproductive status: Female patients of childbearing age or male patients whose sexual partners are female patients of childbearing age are willing to take medically approved and highly effective contraceptive measures , such as intrauterine devices or condoms, from the time the informed consent is signed until 12 months after cell infusion (female patients of childbearing age include premenopausal women and women within 24 months of postmenopause).
10. The subjects must sign and date the written informed consent form.
11. Subjects must be willing and able to comply with the scheduled treatment regimen, laboratory tests, follow-up and other study requirements.

Exclusion Criteria:

1. Pregnant and breastfeeding women.
2. Positive human immunodeficiency virus (HIV) antibody test; hepatitis B virus infection ( HBsAg positive and/or HBc antibody positive, and HBV-DNA positive ); acute or chronic active hepatitis C (HCV antibody positive and HCV-RNA positive ); positive syphilis antibody test; Epstein-Barr virus infection (IgM positive); cytomegalovirus (CMV) infection (IgM positive) ; human T- lymphotropic virus ( HTLV ) positive; positive for novel coronavirus (COVID-19) and not reverting to negative within 7 days . The above pathogen test results are subject to the central laboratory test results.
3. Known HER2 expression is positive (defined as IHC 3+, or IHC 2+ and FISH+).
4. Active or clinically poorly controlled serious infection.
5. Patients had uncontrollable pleural effusion, pericardial effusion, and ascites before enrollment.
6. Extensive or diffuse lung metastases or extensive or diffuse liver metastases or extensive or diffuse bone metastases .
7. Blood oxygen saturation is ≤ 95% without oxygen inhalation.
8. Other serious pulmonary diseases that may limit their participation in this study, such as pulmonary embolism, chronic obstructive pulmonary disease, symptomatic or poorly controlled interstitial lung disease, or clinically significant abnormalities in pulmonary function tests.
9. Patients with deep and large ulcers of the primary lesion, or recurrence of the anastomotic site with tumor infiltration of the entire layer, or tumor lesions infiltrating large blood vessels, who are judged by the researchers to be at high risk of bleeding or perforation, were included in the CT/MRI or combined gastroscopy examinations.
10. Patients with known past or current hepatic encephalopathy requiring treatment; patients with current or history of central nervous system diseases, such as epileptic seizures, cerebral ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease involving the central nervous system; patients with clinical symptoms of central nervous system metastasis or meningeal metastasis, or other evidence indicating that the patient's central nervous system metastasis or meningeal metastasis has not been controlled, who are judged by the investigator to be unsuitable for inclusion.
11. unstable heart disease that requires treatment or heart disease that cannot be controlled after treatment, or hypertension that is poorly controlled as determined by the researchers (defined as systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure > 100 mmHg after standard antihypertensive drug treatment); or diabetes that is still poorly controlled after standard treatment (fasting blood glucose ≥ 10.2 mmol/L).
12. Any of the following cardiac clinical symptoms or diseases within 6 months before cell infusion:

    1. Left ventricular ejection fraction (LVEF) < 50%;
    2. Myocardial infarction within 1 year; or unstable angina; or history of percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG); use of pacemaker;
    3. Resting electrocardiogram (ECG) with QTc F >450 ms (male) or QTc F >470 ms (female);
    4. Resting electrocardiogram reveals clinically significant abnormalities (such as abnormalities in heart rate, conduction, or morphological characteristics), complete left bundle branch block, third- degree atrioventricular block, or a PR interval greater than 250 ms.
13. Evidence of a significant coagulopathy or other significant bleeding risk, including:

    1. clinically significant coagulation abnormalities;
    2. A history of intracranial hemorrhage or spinal cord hemorrhage;
    3. Patients whose tumor lesions invade large blood vessels and have a significant risk of bleeding;
    4. Patients with current unstable or active ulcers or active gastrointestinal bleeding;
    5. An embolic event occurred within 6 months before cell transfusion;
    6. Clinically significant hemoptysis or significant bleeding in tumor lesions occurred within 1 month before cell transfusion;
    7. Major trauma or major surgery within 1 month before enrollment;
    8. The presence of any bleeding disorders, such as hemophilia, von Willebrand disease, etc.;
    9. Use of anticoagulant therapy (except low molecular weight heparin) for therapeutic purposes within 2 weeks before cell transfusion;
    10. Patients are currently receiving conventional anticoagulant therapy (such as warfarin or heparin). Patients require long-term antiplatelet therapy (aspirin ≥ 100 mg/day; clopidogrel ≥ 75 mg/day); dipyridamole, ticlopidine, or cilostazol.
14. Receipt of systemic steroids equivalent to >15 mg/day of prednisone for more than 3 days within 2 weeks before apheresis, excluding inhaled steroids.
15. Subjects requiring systemic treatment with corticosteroids or other immunosuppressive drugs during treatment. Subjects with any active autoimmune disease, or a history of autoimmune disease with expected recurrence (including but not limited to systemic lupus erythematosus, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, and asthma requiring medical intervention with bronchodilators). Exceptions include: type 1 diabetes; skin diseases not requiring systemic treatment (e.g., vitiligo, psoriasis); alopecia; hypothyroidism requiring only hormone replacement therapy; asthma that fully resolved in childhood and does not require any intervention in adulthood; or other subjects whose condition is not expected to relapse in the absence of external triggers.
16. Patients with previous or concurrent malignancies, with the following exceptions:

    1. Adequately treated basal cell or squamous cell carcinoma of the skin (adequate wound healing was required before study enrollment);
    2. Carcinoma in situ of cervical or breast cancer who has undergone curative treatment and has no signs of recurrence for at least 3 years before the study;
    3. The primary malignancy has been completely resected and remains in complete remission for ≥ 5 years.
17. Subjects who have previously received other gene therapies, including but not limited to CAR-T therapy and TCR-T therapy .
18. Received the following treatments or drugs before cell infusion: received chemotherapy, targeted therapy, biological therapy, endocrine therapy, immunotherapy and other anti-tumor treatments (except for treatments used in accordance with the protocol requirements before infusion, such as lymphoproliferative conditioning and bridging therapy) , less than 28 days or less than 5 half-lives (whichever is shorter) from the first infusion of treatment in this study ; received traditional Chinese medicine treatment with anti-tumor indications within 2 weeks before cell infusion.
19. There is a history of other severe allergies such as anaphylactic shock.
20. Subjects with severe mental disorders.
21. If a subject develops a new arrhythmia, including but not limited to arrhythmias that cannot be controlled with medication; hypotension requiring pressor medication; or bacterial, fungal, or viral infection requiring intravenous antibiotics , the investigator may determine that the subject is unsuitable for participation in the trial . Subjects who are taking antibiotics to prevent infection may continue to participate in the trial at the investigator's discretion.
22. Participation in other interventional clinical studies and use of study drug within 1 month before the planned IMC 002 infusion .
23. The investigator assesses that the subject is unable or unwilling to comply with the requirements of the study protocol.
24. 4 weeks before the planned apheresis time or plan to receive a live attenuated vaccine during the study.
25. Subjects with gastrointestinal obstruction or obstructive jaundice are deemed unsuitable for participation in this trial by the investigator .
26. Subjects with any other concurrent serious and/or uncontrolled medical conditions who are deemed unsuitable for participation in this trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 96 week
  Progression-Free Survival (PFS)

SECONDARY OUTCOMES:
OS | From the date of randomization until death from any cause, assessed up to 96 weeks.
  Overall survival (OS)

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-09-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT07103668/Prot_001.pdf